CLINICAL TRIAL: NCT03812874
Title: Phase I/II Study of PTX-9908 Injection As an Inhibitor of Cancer Progression in Patients with Non-resectable Hepatocellular Carcinoma Following Transarterial Chemoembolization Treatment
Brief Title: A Study of PTX-9908 Injection for Non-resectable HCC with TACE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TCM Biotech International Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTX-9908-HCC-01
Record Dates: First submitted 2019-01-15; First posted 2019-01-23 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Phase I: Singe-arm, open-labeled Phase II: Randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For Phase II only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTX-9908 Injection group (Experimental): IV injection.
  Interventions: Drug: PTX-9908 Injection
- Placebo/Vehicle group (Placebo Comparator): IV injection
  Interventions: Drug: PTX-9908 Injection; Drug: Placebo

INTERVENTIONS:
Drug: PTX-9908 Injection — Proposed dose cohorts:1 mg/kg, 2 mg/kg, 4 mg/kg, 8 mg/kg, and 16 mg/kg.
  Frequency:
  Phase I: one dose per day for 4 consecutive weeks (20 doses). Phase II (A)Daily Dose Regimen one dose per day for 12 consecutive weeks (60 doses). (B) Daily for first week, followed by weekly treatment Regimen One dose per day for 5 consecutive days in Week 1 (5 doses), and one dose per week till for 11 weeks (11 doses).
  Duration: 4 weeks (Phase I) and 12 weeks (Phase II).
Drug: Placebo — water for injection
  Phase II (A)Daily Dose Regimen one dose per day for 12 consecutive weeks (60 doses). (B) Daily for first week, followed by weekly treatment Regimen One dose per day for 5 consecutive days in Week 1 (5 doses), and one dose per week till for 11 weeks (11 doses).
  Duration: 12 weeks (Phase II)
  Arms: Placebo/Vehicle group

SUMMARY:
This is a multicenter, Phase I/II study in patients with non-resectable hepatocellular carcinoma following TACE treatment.

Phase I (Open-label dose escalation)

This study will be an open-label study with an Accelerated Phase and a Standard Phase. For the Accelerated Phase of the study, one patient per dose level (1 mg/kg, and 2 mg/kg) is planned. For the dose levels in the standard phase (4 mg/kg, 8 mg/kg and 16 mg/kg), it will follow the Fibonacci's rule of 3 + 3 design. All eligible patients who have received TACE treatment and recovered well, will be administrated PTX-9908 Injection intravenously one dose per day for 5 days on Week 1 (excludes weekends and public holidays), and one dose per week (on Day 8, Day 15, and Day 22) for 3 consecutive weeks. The 4-week treatment period, will be followed by a 2-week follow-up period.

Phase II (Randomized placebo controlled dose expansion)

The objective of phase II is to further evaluate the safety, tolerability and antitumor activity of PTX-9908 Injection for patients with non-resectable hepatocellular carcinoma following TACE treatment. Approximately 24 eligible patients who have received TACE treatment and recovered, will be randomized to PTX-9908 Injection using the predetermined dose in phase I or the vehicle placebo in a 2:1 ratio. PTX-9908 Injection or placebo will be administered intravenously one dose per day for 5 days in Week 1 (excludes weekends and public holidays), and one dose per week till Week 12 (Day 78). The 12-week treatment period, will be followed by a 2-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable hepatocellular carcinoma and at intermediate-stage HCC (BCLC stage B or Child-Pugh class A/B with large or multifocal HCC, no vascular invasion, or extrahepatic spread) with completed TACE procedure in 4 weeks before day 1 of study intervention infusion.
2. Recovered from TACE treatment and procedure related toxicities including ALT/AST and bilirubin within normal limit or reference numeric value (reference value is defined as the test value before TACE procedure).
3. ECOG (Eastern Cooperative Oncology Group) performance status < 2.
4. Have adequate organ and marrow function as defined below:

   1. Absolute neutrophil count > 1,200/µL
   2. Hemoglobin > 9 g/dL
   3. Platelets > 100,000/µL
   4. Total bilirubin < 2 X ULN
5. Have adequate kidney function as estimated glomerular filtration rate (eGFR) > 60 mL/min/1.73m2
6. A negative pregnancy test at screening. This applies to any female patient with childbearing potential.
7. Agree to use adequate contraception after signing informed consent form, during the duration of study participation and for at least 4-weeks after completion or withdrawal from the study. This applies to any female patient with childbearing potential and any male patient whose female partner has childbearing potential.

   Acceptable contraceptive methods include:
   1. Established use of oral, injected or implanted hormonal methods of contraception
   2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
   3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) >=20 years of age. (Note: In Taiwan, age of majority recognized in law is 20 years of age)
8. >=20 years of age. (Note: In Taiwan, age of majority recognized in law is 20 years of age)
9. Anticipated life expectancy of >= 6 months at assessment during screening.
10. Ability to understand and have signed a written informed consent document.

Exclusion Criteria:

1. 1. Patient with Child-Pugh B8-9.
2. Patient who has had anti-cancer therapy including surgery, radiotherapy, immunotherapy, or chemotherapy (except in TACE regimen) within 4 weeks prior to the screening visit.
3. Patient who has received any other investigational agents within 4 weeks prior to the screening visit.
4. Patient who has not recovered from the side effects of the earlier investigational agent or had anti-cancer therapy including surgery, radiotherapy, immunotherapy, or chemotherapy.
5. Patient with known brain metastases, leptomeningeal or epidural metastases (unless treated and well controlled for >= 3 months).
6. Patient with prior history of co-malignancies, except for adequately treated carcinoma in situ of the cervix, ductal carcinoma in situ (DCIS) of the breast, and basal cell/squamous cell skin cancer.
7. Patient with history of myocardial infarction or uncontrolled cardiac dysfunction, or unstable arrhythmia or symptomatic peripheral arterial vascular disease.
8. Patient with history of positive serology for human immunodeficiency virus (HIV).
9. Patient with active, uncontrolled bacterial, viral, or fungal infections, which require systemic therapy.
10. Patient with poor liver function as indicated by serum bilirubin > 2 mg/dL, Child-Pugh Class C, severe coagulopathy (INR > 2) not correctable with vitamin K, or active hepatic encephalopathy.
11. Patient with known allergic reactions to biological agent or polypeptides similar to PTX-9908 Injection.
12. Woman who is pregnant or nursing.
13. Patient with concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the patient in this study.
14. Patient with unwillingness or inability to comply with the study protocol for any reason.
15. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE grade 1) using Frederica's QT correction formula
16. A history of additional risk factors for torsades de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
17. The use of concomitant medications that prolong the QT/QTc interval

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-10-06 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by the number and severity of Adverse Events | Week 1 - Week 8 (Phase I)/Week 16 (Phase II)
Safety as measured by number of participants with a dose limiting toxicity (DLT) | Week 1 - Week 6 (Phase I only)
  Any of the following, if judged to be associated with PTX-9908 Injection or the combination of TACE with PTX-9908 Injection (i.e., with possible causality) that occur within the DLT evaluation window, will be considered as a DLT.
  1. All Grade 4 (i.e., life-threatening) non-hematological and hematological toxicities (except for Grade 4 lymphopenia).
  2. Grade 3 anemia with clinically significant bleeding
  3. All grades of febrile neutropenia.
  4. All Grade 3 non-laboratory/non-hematologic treatment-emergent adverse events, with the exception for nausea, vomiting, or diarrhea that resolves within 3 days.
  5. Grade 3 thrombocytopenia with clinically significant bleeding is a DLT.
  6. Grade 3 cytokine release syndrome of any duration is a DLT.
  7. Grade 3 laboratory adverse events that are judged by the investigator as clinically significant.

SECONDARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Week 1 - Week 6 (Phase I only)
  The RP2D was based on the highest dose in which 0/6 or 1/6 participants experienced DLT with at least 2 out of no more than 6 participants experiencing DLT at the next higher dose level, and the assessment of any relevant chronic toxicity.
Maximum Plasma Concentration (Cmax) of single-dose and repeat-dose of PTX-9908 Injection | Day 1, Day 5, Day 8, Day 15, and Day 26 in Phase I and Phase II
  Pharmacokinetics (PK) is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. Cmax=maximum observed plasma concentration of PTX-9908 Injection administered with IV dose derived from plasma concentration versus time data.
Terminal Half-life (T-Half) of single-dose and repeat-dose of PTX-9908 Injection | Day 1, Day 5, Day 8, Day 15, and Day 26 in Phase I and Phase II
  PK is a branch of pharmacology concerned with the rate at which drugs are absorbed, distributed, metabolized, and eliminated by the body. T-Half=terminal-phase elimination half-life in plasma of PTX-9908 Injection administered with IV.
Overall Tumor Response | Week 1 - Week 16 (Phase II)
  Number of participants with a best overall tumor response of complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD). Overall tumor response will be assessed using contrast-enhanced CT imaging according to mRECIST criteria following the 1.1 release of RECIST.
Response of target hepatic lesions in embolized territory | Week 1 - Week 16 (Phase II)
  Number of participants with hepatic lesion in embolized territory of complete Response (CR), Partial Response (PR), Stable Disease (SD), and Progressive Disease (PD). Tumor response will be assessed using contrast-enhanced CT imaging according to mRECIST criteria following the 1.1 release of RECIST
To evaluate overall time-to-progression | Week 1 - Week 16 (Phase II)
  Time to progression (TPP) will start from TACE administration to radiological progression. Definition of progression is based on the mRECIST criteria.
To evaluate change in AFP levels. | Week 1 - Week 16 (Phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Hung Chien-Hung, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, New Taipei City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided